CLINICAL TRIAL: NCT01681693
Title: Effect of Genetic Variants in MATE1 and OCT3 Transporters on the Pharmacodynamics of Metformin in African Americans With Type II Diabetes Mellitus.
Brief Title: Effect of Genetic Variants in MATE1 and OCT3 on the Pharmacodynamics of Metformin in African Americans
Acronym: #6113
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6113
Record Dates: First submitted 2012-08-01; First posted 2012-09-10 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Healthy; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): Subjects will be given an oral dose of metformin once per day for two days.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Subjects will be given an oral dose of metformin once per day for two days.
  Other Names: GLUCOPHAGE

SUMMARY:
The current study is part of a large multi-investigator grant to look at the pharmacogenetics of a number of membrane transporters. The investigators will study individuals with particular genotypes of the human organic cation transporter, (hOCT3), and the multidrug and toxin extrusion transporter, MATE1 to test the hypothesis that genetic variation in hOCT3 and hMATE1 are associated with variation in the pharmacokinetics and/or pharmacodynamics of the antidiabetic agent, metformin.

DETAILED DESCRIPTION:
To investigate the potential association of polymorphic genetic variants MATE1 and OCT3 with altered response to metformin, a genotype to phenotype strategy is employed. Specifically, the investigators will evaluate this hypothesis in African-Americans, a population which has a high incidence of type 2 diabetes and which has high variant allele frequencies (44.5% for MATE1-66T>C and 11.3% in OCT3-81G>delGA) relative to other ethic groups. To assess the effects of these variants on metformin response, the investigators will measure metformin renal clearance (pharmacokinetics of metformin), and plasma glucose and insulin levels (pharmacodynamic response) in healthy and diabetic patients who carry either the reference or variant alleles.

ELIGIBILITY:
Inclusion Criteria:

* Subjects self-identify racial background, identify themselves, parents and four grandparents as African American
* Subject status is healthy volunteer from t In the event that diabetes is indicated in a normal subject based on OGTT results, we will notify the patients' primary care physician. he SOPHIE cohort OR diagnosis of T2DM based on American Diabetes Association (ADA) criteria
* Subjects over 18 years old and below 60 years
* Subjects who are healthy on the basis of medical history, physical examinations and laboratory tests if healthy volunteer from SOPHIE
* Subjects who agree with the written informed consent to participate in the study

Exclusion Criteria:

* Unable to confirm African-American ethnicity
* Under 18 years old
* Pregnant or lactating women (female subjects will have a urine pregnancy test at the screening visit).
* Prior history of any allergic reaction to metformin
* Has a risk of congestive heart failure requiring pharmacologic treatment (medical history)
* Has a prior history of renal* or hepatic dysfunction (renal and hepatic function will be evaluated based on screening blood tests conducted prior to study enrollment)
* Risk of urinary or gastric retention or narrow-angle glaucoma (by medical history examination)
* Impaired renal function (e.g as suggested by abnormal creatinine clearance, eGFR <60 or serum creatinine >1.4 mg/dl in females and >1.5 mg/dl in males) which may also result from conditions such as cardiovascular collapse (shock), acute myocardial infarction (heart attack), and septicemia, abnormal heart rhythms (tachyarrhythmias; heart beat > 100 beats per minute).
* Impaired hepatic function (> 1.5 times the upper limit of normal)
* Evidence of anemia (hemoglobin <10 g)
* Taking a medication that could confound study results, such as known substrates or inhibitors of OCT3 and MATE1, such as cimetidine.
* They do not provide consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Renal Clearance of the Metformin | 24 hours post-dose
  To test whether individuals with genetic variants of transporters OCT3 and MATE1 exhibit altered pharmacokinetics of metformin.
Plasma glucose | 0, 15, 30, 45, 60, 90, 120, 180 minutes after glucose administration
  To test whether individuals with genetic variants of transporters OCT3 and MATE1 exhibit altered glucose lowering response to metformin.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Giacomini, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States